CLINICAL TRIAL: NCT02135185
Title: Phase II Study, Multicentric, Randomized Studying the Effect of the Rehabilitation Effort at Home in Patients With Head and Neck Tumor Treated With Curative Intent
Brief Title: Effect of the Rehabilitation Effort at Home in Patients With Head and Neck Tumor Treated With Curative Intent
Acronym: NUTRIMOUV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VA2011/43
Record Dates: First submitted 2014-02-06; First posted 2014-05-09 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rehabilitation effort (Experimental): custom work endurance combining dietary management adapted to the nutritional status and an APA. Included patients benefit from support for 19 weeks from the start of treatment
  Interventions: Other: custom work endurance
- Control (Active Comparator): Control with dietary management adapted to the nutritional status
  Interventions: Behavioral: dietary management adapted to the nutritional status

INTERVENTIONS:
Other: custom work endurance — Experimental: Rehabilitation effort
  Arms: Rehabilitation effort
Behavioral: dietary management adapted to the nutritional status — dietary management adapted to the nutritional status
  Arms: Control

SUMMARY:
Improvement exercise tolerance

DETAILED DESCRIPTION:
This study allows improved exercise tolerance in patients undergoing rehabilitation effort

ELIGIBILITY:
Inclusion Criteria:

* Tumor squamous cell head and neck (excluding nasopharynx) nonmetastatic including cervical lymphadenopathy primitives
* Patient to be treated with curative radiotherapy monofractionnée for at least 6 weeks, with or without concurrent chemotherapy (including targeted therapies)
* KPS ≥ 60

Exclusion Criteria:

* Cancer of the nasopharynx
* Metastatic Patient
* Patients who received neoadjuvant chemotherapy or induction
* Patient parenteral nutrition
* Non-compliant Patient Treatment
* Patient with a cons-indication to the achievement of an effort: clinical signs of pulmonary arterial hypertension (PAH) uncontrolled heart failure, recent myocardial infarction, arrhythmias, unstable angina.
* Patient desaturation in the stress test
* Patient already included in another clinical trial with an experimental molecule
* Pacemaker or defibrillator or neurostimulator
* Contraindications to treatment with standard radiotherapy with or without concurrent chemotherapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
measurement of the increase of initial endurance | up to 24 weeks
  Patients increasing rate of at least 40% of their initial endurance time 3 months after the completion of radiotherapy

SECONDARY OUTCOMES:
Quality of life | 3 months after the end of radiotherapy
  Quality of life 3 months after the end of radiotherapy (QLQ C30 and SF 36)
Quality of life | 3 months after the end of radiotherapy
  "Performance status" (Karnofsky) 3 months after the end of radiotherapy.
Quality of life | 3 months after the end of radiotherapy
  Quantity of daily physical activity to 3 months after the end of radiotherapy (Actimeter).
Quality of life | 3 months after the end of radiotherapy
  Decrease addiction to 3 months after the end of radiotherapy (Declarative).
Quality of life | 3 months after the end of radiotherapy
  Rate of feasibility of the protocol.
Quality of life | 3 months after the end of radiotherapy
  Identification of indicator (s) to monitor the APA.
Quality of life | 3 months after the end of radiotherapy
  Evaluation of precariousness (EPICES).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SENESSE, Principal Investigator — ICM Co. Ltd.
Locations (1):
- Institut régional du Cancer - Montpellier - Val d'Aurelle, Montpellier, France

REFERENCES:
- [Derived] Vinches M, Janiszewski C, Thezenas S, Delample D, Boisselier P, Jacquot S, Senesse P, Faravel K. Evaluation of physical rehabilitation in patients receiving curative treatment for head and neck cancer: The NUTRIMOUV randomized phase II trial. Support Care Cancer. 2025 Dec 16;34(1):35. doi: 10.1007/s00520-025-10265-7. PMID 41400716